CLINICAL TRIAL: NCT03167632
Title: Oral Ulcer Prevalence of and Quality of Life: a Hospital-based Cross-sectional Study
Brief Title: Oral Ulcer Prevalence: Hospital-based Cross-sectional Study
Status: Completed | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ayat Gamal-AbdelNaser, Teaching assistant, Cairo University
Other Study IDs: QoL1
Record Dates: First submitted 2017-05-24; First posted 2017-05-30 (Actual); Last update posted 2017-05-30 (Actual); Status verified 2017-05

CONDITIONS: Oral Ulcer
MeSH Terms: conditions — Oral Ulcer

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- dental patients

SUMMARY:
Oral Ulcers have serious effect on patients' lives. Due to absence of any information about its prevalence, risk factors and effect on patients' lives, this study has been held. The investigators recruited patients from the outpatient dental clinic of the faculty of oral and dental medicine, Cairo University, screened them clinically for oral ulcers. All patients filled questionnaires about the risk factors of oral ulcers. Furthermore, oral ulcer patients filled questionnaires about their Quality of life, previous treatments used, previous physicians visited and their Quality of life after using previous treatments.

DETAILED DESCRIPTION:
Oral ulcers form a category of oral lesions that is frequently encountered by the dentist. It influences the patients' lives greatly. In a first step to reducing the disease burdens on patients, basic data about the disease distribution and possible risk factors should be gathered through epidemiological studies.

This cross-sectional study consisted of a convenience sample of 605 dental patients recruited in the time from August to October 2015. The study was held in the outpatient oral diagnosis clinic, Faculty of Oral and Dental Medicine, Cairo University, Egypt; which is an open public facility, a tertiary healthcare and a referral center.

For each participant, the study details were explained and the consent was received. Then, medical history was taken, comprehensive oral examination was done, history of any detected oral ulcer was investigated. The questionnaire was filled through a face-to-face interview.

Comprehensive oral examination was held on a dental unit using the light of the unit, mirror and probe.

After full examination and questionnaire filling, the oral ulcer patients were educated about their oral problem and their ulcers were managed. If the patient's condition needed further investigations or management, referral was done to the appropriate department of the faculty.

The Questionnaire included a section for demographic information of age, sex, social and educational levels of the patient. It also included questions about medical condition, habits of trauma, smoking and its frequency.

After examination, if an ulcer was detected, a part of the questionnaire was filled describing the ulcer: site, size, number, shape, distribution, depth, edges, floor, margins, induration and regional lymph node status. Also, the (OHIP-14) questionnaire was filled to assess the effect of the ulcer on the patient's quality of life.

The questionnaire included questions about previous treatments used by the patients, the patients' assessment of their effect and the source of the patients' information about these therapies.

The patients was also asked about their previous experiences with dentists or physicians seeked to treat these ulcers.

ELIGIBILITY:
Inclusion Criteria:

* Subjects whose age was above 15 years old.

Exclusion Criteria:

* Subjects having problem in opening their mouth (due to non-oral ulcer cause) or undergoing intermaxillary fixation where oral examination was not possible.

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: patients attending the outpatient clinic of oral diagnosis, department of Oral Medicine, Oral Diagnosis and Periodontology, Faculty of Oral and Dental Medicine, Cairo University.
Sampling Method: Non-Probability Sample
Enrollment: 605 (Actual)
Dates: Start 2015-08-10 (Actual); Primary Completion 2015-10-25 (Actual); Study Completion 2015-10-25 (Actual)

PRIMARY OUTCOMES:
prevalence of Oral Ulcers | 3 months
  number of patients having oral ulcers

SECONDARY OUTCOMES:
Oral health related-quality of life (OHR-QoL). | 3 months
  Quality of life of patients having oral ulcers
The effect of previous treatment | 3 months
  measured by: OHIP-14 at the end of treatment and the time interval of ulcer-free period after stoppage of treatment.
Types of non-conventional treatments used | 3 months
  reported together with its side effects as nominal outcomes.
Number of dentists or physicians visited before | 3 months
  Also the specialties of these physicians reported

IPD SHARING:
Plan to Share IPD: Yes
Whenever asked for meta-analysis, the IPD will be available in the form of an excel sheet having no identifiers, where each patient is given an ID number of the study.